CLINICAL TRIAL: NCT00448136
Title: An Open Label Study to Evaluate the Effect of Avastin in Association With Chemotherapy on Progression-free Survival in Patients With Progressive Advanced/Metastatic Well-differentiated Digestive Endocrine Tumors of the Gastrointestinal Tract
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Chemotherapy in Patients With Endocrine Tumors of the Gastrointestinal Tract.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20383
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab; Streptozocin; Capecitabine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: 5 FU; Drug: Streptozotocin
- 2 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Xeloda

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg iv on day 1 every 3 weeks
Drug: 5 FU — 400mg/m2/day iv on days 1-5 every 6 weeks
  Arms: 1
Drug: Streptozotocin — 500mg/m2/day iv on days 1-5 every 6 weeks
  Arms: 1
Drug: Xeloda — 1000mg/m2 po bid on days 1-14 every 3 weeks
  Arms: 2

SUMMARY:
This 2 arm study will assess the efficacy and safety of two systemic treatments including Avastin in patients with previously-untreated progressive locally advanced/metastatic well-differentiated digestive endocrine tumors. Patients with duodeno-pancreatic tumors (arm 1) will be treated with 5FU/streptozotocin iv (5FU 400mg/m2/d D1 to D5;streptozotocin 500mg/m2/d/iv D1 to D5;D1=D42) every 6 weeks, plus Avastin 7.5mg/kg iv every 3 weeks. Patients with gastrointestinal tract tumors (arm 2) will be treated with Xeloda 1000mg/m2 po bid D1 to D14 plus Avastin 7.5mg/kg iv D1=D21 every 3 weeks. The patients will be treated with chemotherapy for a minimum of 6 months, unless there is tumor progression and/or unacceptable toxicity. The anticipated time on study treatment is until disease progression or unacceptable toxicity, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* well-differentiated gastrointestinal tract endocrine tumors, or duodeno-pancreatic endocrine tumors;
* no previous anti-cancer therapy, other than surgery;
* progressive metastatic disease;
* >=1 measurable lesion.

Exclusion Criteria:

* abnormal cardiac function, with history of ischemic heart disease in past 6 months and/or abnormal 12 lead ECG;
* patients with known bleeding disorders;
* unstable systemic disease;
* chronic daily treatment with high-dose aspirin, NSAIDs or corticosteroids;
* previous history of malignancy (other than successfully treated basal and squamous cell cancer of the skin, and/or in situ cancer of the cervix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- France (22):
  - Angers
  - Bordeaux
  - Boulogne-Billancourt
  - Caen
  - Chambray-lès-Tours
  - Clichy
  - Créteil
  - Dijon
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Poitiers
  - Reims
  - Rouen
  - Saint-Brieuc
  - Strasbourg
  - Toulouse
  - Villejuif

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + 5-fluorouracil (5-FU) + Streptozocin: Cycles 1-5 (42-day cycles): Participants received bevacizumab 7.5 milligrams per kilogram (mg/kg) intravenously (IV) on Days 1 and 22; 5-FU 400 mg per square meter per day (mg/m^2/day) IV on Days 1 through 5; and streptozocin 500 mg/m^2/day IV on Days 1 through 5. Days 5-21 and 23-42 were rest periods. This 42-day cycle was repeated at least 4 times.
- Bevacizumab + Capecitabine: Cycles 1-9 (21-day cycles): Participants received bevacizumab 7.5 mg/kg IV on Day 1; capecitabine 1000 mg/m^2, tablets, orally (PO), twice daily (BID) on Days 1 through 14. Days 15-21 were a rest period. This 21-day cycle was repeated at least 8 times.
Period: Overall Study
Arm/Group | Bevacizumab + 5-fluorouracil (5-FU) + Streptozocin | Bevacizumab + Capecitabine
Started | 34 | 49
Completed | 30 | 41
Not Completed | 4 | 8
Not completed — Death | 3 | 8
Not completed — Investigator's decision (progression) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of treatment.
Groups:
- Bevacizumab + 5-FU + Streptozocin: Cycles 1-5 (42-day cycles): Participants received bevacizumab 7.5 mg/kg IV on Days 1 and 22; 5-FU 400 mg/m^2/day IV on Days 1 through 5; and streptozocin 500 mg/m^2/day IV on Days 1 through 5. Days 5-21 and 23-42 were rest periods. This 42-day cycle was repeated at least 4 times.
- Bevacizumab + Capecitabine: Cycles 1-9 (21-day cycles): Participants received bevacizumab 7.5 mg/kg IV on Day 1; capecitabine 1000 mg/m^2, tablets, PO, BID on Days 1 through 14. Days 15-21 were a rest period. This 21-day cycle was repeated at least 8 times.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine | Total
Number analyzed (Participants) | 34 | 49 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.93 (10.63) | 61.64 (9.20) | 59.29 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 23 | 35
  Male | 22 | 26 | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS is defined as the interval between the date of start of treatment and the date of evaluation by the investigator of progressive disease or death from any cause. The progression was assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) using medical imaging during the treatment period and by the investigators (confirmed by medical imaging) during the follow-up period. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of disease progression or death were censored at the date of the last visit or follow-up without progression.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 49
percentage of participants | 52.9 | 53.1

2. Secondary Outcome: Percentage of Participants With a Response by Best Overall Response
Description: Best overall response defined as best response recorded during the study as defined according to RECIST; performed by the investigator and by centralized review. Complete response (CR): complete disappearance of all target lesions and non-target disease. All lesions, both target and non-target, must have decreased to normal (short axis, less than [<]10 millimeters [mm]). No new lesions. Partial response (PR): greater than or equal to (≥)30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter (LD) was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Stable disease (SD): not qualifying for CR, PR, or Progressive Disease (PD). PD: at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population. Data were missing from centralized review for 1 participant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 49
percentage of participants
  PR (Investigator) | 55.9 [39.2 to 72.6] | 18.4 [7.5 to 29.2]
  PR (Centralized review) | 51.5 [34.5 to 68.6] | 12.5 [3.1 to 21.9]
  SD (Investigator) | 44.1 [27.4 to 60.8] | 69.4 [56.5 to 82.3]
  SD (Centralized review) | 48.5 [31.4 to 65.5] | 81.3 [70.2 to 92.3]
  PD (Investigator) | 0 [0 to 0] | 8.2 [0.5 to 15.8]
  PD (Centralized review) | 0 [0 to 0] | 0 [0 to 0]
  Not evaluable (Investigator) | 0 [0 to 0] | 4.1 [0.0 to 9.6]
  Not evaluable (Centralized review) | 0 [0 to 0] | 6.3 [0.0 to 13.1]

3. Secondary Outcome: Duration of Overall Response (OR) - Percentage of Participants With an Event
Description: Determined only for those participants with an overall response (CR or PR) and was defined as the time interval between the response (CR or PR) and the date of progression or death from any cause. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of progression or death were censored at the data of last visit or follow-up without progression.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population; only participants with a response of CR or PR were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 19 | 9
percentage of participants | 42.1 | 22.2

4. Primary Outcome: PFS - Time to Event
Description: PFS is defined as the interval between the date of start of treatment and the date of evaluation by the investigator of progressive disease or death from any cause. The progression was assessed according to RECIST using medical imaging during the treatment period and by the investigators (confirmed by medical imaging) during the follow-up period. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of disease progression or death were censored at the date of the last visit or follow-up without progression. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 49
months | 23.7 [13.1 to NA] — The upper limit for the median PFS was not estimated because it was longer than the latest censoring time, and therefore was not achieved. | 23.4 [13.2 to NA] — The upper limit for the median PFS was not estimated because it was longer than the latest censoring time, and therefore was not achieved.

5. Primary Outcome: PFS - Percentage of Participants Estimated to be Progression Free at 12 and 24 Months
Description: PFS is defined as the interval between the date of start of treatment and the date of evaluation by the investigator of progressive disease or death from any cause. The progression was assessed according to RECIST using medical imaging during the treatment period and by the investigators (confirmed by medical imaging) during the follow-up period. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of disease progression or death were censored at the date of the last visit or follow-up without progression.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 49
percentage of participants
  12 months | 76 | 65
  24 months | 50 | 48

6. Secondary Outcome: Duration of OR - Time to Event
Description: Determined only for those participants with an overall response (CR or PR) and was defined as the time interval between the response (CR or PR) and the date of progression or death from any cause. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of progression or death were censored at the data of last visit or follow-up without progression. Median duration of OR was estimated using the Kaplan-Meier method.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population; only participants with a response of CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 19 | 9
months | NA [11.2 to NA] — Median duration and upper limit of the 95% confidence interval (CI) could not be calculated due to an insufficient number of events. | NA [3.2 to NA] — Median duration and upper limit of the 95% CI could not be calculated due to an insufficient number of events.

7. Secondary Outcome: Duration of OR - Percentage of Participants With Sustained Response at 12 and 24 Months
Description: Duration of OR was determined only for those participants with an overall response of CR or PR and was defined as the time interval between the response (CR or PR) and the date of progression or death from any cause. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of progression or death were censored at the data of last visit or follow-up without progression.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 19 | 9
percentage of participants
  12 months | 74 | 70
  24 months | 55 | NA — Not evaluable as data from all participants were censored, or participants had experienced events of progression or death before the 24-month timepoint.

8. Secondary Outcome: Duration of Overall Disease Control (ODC) - Percentage of Participants With an Event
Description: Determined only for those participants with overall disease control (CR, PR or SD per RECIST) and was defined as the time interval between the first occurrence of disease control (CR, PR or SD) and the date of progression or death from any cause. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of progression or death were censored at the data of last visit or follow-up without progression.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 43
percentage of participants | 52.9 | 46.5

9. Secondary Outcome: Duration of ODC - Time to Event
Description: Determined only for those participants with overall control disease (CR, PR, or SD per RECIST) and was defined as the time interval between the first occurrence of disease control (CR, PR or SD) and the date of progression or death from any cause. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of progression or death were censored at the data of last visit or follow-up without progression. Median time to event was estimated using the Kaplan-Meier method.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population; only participants with a response (CR, PR, or SD) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 43
months | 22.3 [11.9 to NA] — The upper limit of the 95% CI was not estimated because it was longer than the latest censoring time, and therefore was not achieved. | 23.4 [15.1 to NA] — The upper limit of the 95% CI was not estimated because it was longer than the latest censoring time, and therefore was not achieved.

10. Secondary Outcome: Duration of ODC - Percentage of Participants Maintaining Disease Control at 12 and 24 Months
Description: Duration of ODC was determined only for those participants with overall control disease (CR, PR, or SD per RECIST) and was defined as the time interval between the first occurrence of disease control (CR, PR, or SD) and the date of progression or death from any cause. Data for participants who were lost to follow-up were censored at the date of last evaluation without progression. Data for participants who completed the study without an event of progression or death were censored at the data of last visit or follow-up without progression.
Time Frame: Screening, every 3 months during treatment, every 6 months during follow-up to 2 years
Population: ITT population; only participants with a response (CR, PR, or SD) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 43
percentage of participants
  12 months | 68 | 72
  24 months | 42 | NA — Not evaluable as data from all participants were censored, or participants had experienced events of progression or death before the 24-month timepoint.

11. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the first treatment administration to death from any cause. Data for participants who were lost to follow-up were censored at the date of last evaluation. Data for participants who were alive at the end of the study were censored at the date of last visit.
Time Frame: Screening, Day 1 of every cycle during treatment, every 6 months during follow-up to 2 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 49
percentage of participants | 14.7 | 16.3

12. Secondary Outcome: OS - Time to Event
Description: OS was defined as the time from the first treatment administration to death from any cause. Data for participants who were lost to follow-up were censored at the date of last evaluation. Data for participants who were alive at the end of the study were censored at the date of last visit. Median OS was estimated using the Kaplan-Meier method.
Time Frame: Screening, Day 1 of every cycle during treatment, every 6 months during follow-up to 2 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 49
months | NA [27 to NA] — The median (and upper 95% CI) OS was not estimated because it was longer than the latest censoring time, and therefore was not achieved. | NA [NA to NA] — The median OS was not estimated because it was longer than the latest censoring time, and therefore was not achieved.

13. Secondary Outcome: OS - Percentage of Participants Surviving at 12 and 24 Months
Description: as for outcome 11
Time Frame: Screening, Day 1 of every cycle during treatment, every 6 months during follow-up to 2 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 34 | 49
percentage of participants
  12 months | 94 | 88
  24 months | 88 | 85

14. Secondary Outcome: Global Health Status as Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - C30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores were averaged and transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Screening, every 3 months during treatment
Population: ITT population; only participants who completed the questionnaire at baseline and who had at least 1 post-baseline assessment were included in the analysis. Number (n) equals (=) the number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 29 | 40
units on a scale
  Baseline (n=29,40) | 65.23 (23.89) | 65.42 (20.02)
  3 months (n=20,32) | 65.83 (19.48) | 57.03 (22.41)
  6 months (n=20,24) | 60.00 (21.90) | 66.32 (21.35)
  12 months (n=13,14) | 66.03 (17.83) | 72.62 (19.46)
  End of treatment (n=13,23) | 64.74 (23.36) | 57.97 (28.48)

15. Secondary Outcome: Percentage of Participants With Change From Baseline in Global Health Status by EORTC QLQ-C30 Improvement Category
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms. Changes from baseline were categorized as follows: Very much worsening (less than [<]-20); Moderate worsening (greater than or equal to [≥]-20 to <-10); Little worsening (≥-10 to <-5); No change (≥-5 to less than or equal to [≤]5); Little improvement (>5 to ≤10); Moderate improvement (>10 to ≤20); and Very much improved (>20).
Time Frame: Screening, every 3 months during treatment
Population: ITT population; only participants who completed the questionnaire at baseline and who had at least 1 post-baseline assessment were included in the analysis. n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 20 | 29
percentage of participants
  3 months, Very much worsening (n=20,29) | 10.0 | 17.2
  3 months, Moderate worsening (n=20,29) | 10.0 | 24.1
  3 months, Little worsening (n=20,29) | 10.0 | 17.2
  3 months, No change (n=20,29) | 40.0 | 24.1
  3 months, Little improving (n=20,29) | 5.0 | 3.4
  3 months, Moderate Improving (n=20,29) | 15.0 | 3.4
  3 months, Very much improving (n=20,29) | 10.0 | 10.3
  6 months, Very much worsening (n=20,22) | 15.0 | 22.7
  6 months, Moderate worsening (n=20,22) | 10.0 | 18.2
  6 months, Little worsening (n=20,22) | 5.0 | 0
  6 months, No change (n=20,22) | 35.0 | 31.8
  6 months, Little improving (n=20,22) | 10.0 | 13.6
  6 months, Moderate Improving (n=20,22) | 15.0 | 0
  6 months, Very much improving (n=20,22) | 10.0 | 13.6
  12 months, Very much worsening (n=12,13) | 8.3 | 0
  12 months, Moderate worsening (n=12,13) | 8.3 | 15.4
  12 months - Little worsening (n=12,13) | 33.3 | 15.4
  12 months, No change (n=12,13) | 25.0 | 38.5
  12 months, Little improving (n=12,13) | 8.3 | 7.7
  12 months, Moderate Improving (n=12,13) | 16.7 | 15.4
  12 months, Very much improving (n=12,13) | 0 | 7.7
  End of treatment, Very much worsening (n=13,20) | 15.4 | 15.0
  End of treatment, Moderate worsening (n=13,20) | 30.8 | 5.0
  End of treatment, Little worsening (n=13,20) | 0 | 10.0
  End of treatment, No change (n=13,20) | 15.4 | 45.0
  End of treatment, Little improving (n=13,20) | 15.4 | 10.0
  End of treatment, Moderate Improving (n=13,20) | 15.4 | 5.0
  End of treatment, Very much improving (n=13,20) | 7.7 | 10.0

16. Secondary Outcome: EORTC QLQ-C30 Functional and Symptom Scale Scores
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores averaged, transformed to 0-100 scale; for functional scores, a higher score represents a better level of functioning. For symptom scale scores a higher level represents a more severe level of symptoms.
Time Frame: Screening, every 3 months during treatment
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Number analyzed (Participants) | 30 | 43
units on a scale
  Physical functioning, Baseline (n=30,43) | 90.44 (13.30) | 87.71 (14.88)
  Physical functioning, 3 months (n=22,33) | 89.32 (12.77) | 75.35 (24.07)
  Physical functioning, 6 months (n=21,24) | 81.98 (19.75) | 82.50 (18.21)
  Physical functioning, End of Treatment (n=13,24) | 82.82 (20.21) | 79.44 (19.85)
  Role functioning, Baseline (n=30,43) | 82.22 (27.31) | 83.33 (25.46)
  Role functioning, 3 months (n=22,33) | 85.61 (21.39) | 62.12 (33.66)
  Role functioning, 6 months (n=21,24) | 75.40 (29.16) | 70.83 (28.34)
  Role functioning, End of Treatment (n=13,24) | 78.21 (32.90) | 72.92 (29.00)
  Emotional functioning, Baseline (n=30,42) | 71.94 (28.32) | 71.89 (20.50)
  Emotional functioning, 3 months (n=21,33) | 81.48 (20.53) | 76.01 (24.27)
  Emotional functioning, 6 months (n=21,24) | 72.62 (28.28) | 76.04 (26.27)
  Emotional functioning, End of Treatment (n=13,24) | 77.56 (23.17) | 73.61 (24.04)
  Cognitive functioning, Baseline (n=30,42) | 86.67 (18.26) | 87.30 (16.38)
  Cognitive functioning, 3 months (n=22,33) | 89.39 (15.04) | 83.84 (21.03)
  Cognitive functioning, 6 months (n=21,24) | 83.33 (21.08) | 82.64 (18.04)
  Cognitive functioning, End of Treatment (n=13,24) | 83.33 (22.57) | 81.94 (25.97)
  Social functioning, Baseline (n=30,41) | 86.11 (21.48) | 87.40 (20.34)
  Social functioning, 3 months (n=22,33) | 89.39 (17.48) | 75.76 (27.35)
  Social functioning, 6 months (n=21,24) | 81.75 (26.30) | 83.33 (21.42)
  Social functioning, End of Treatment (n=13,24) | 84.62 (24.96) | 81.94 (21.93)
  Fatigue, Baseline (n=30,42) | 26.30 (23.61) | 27.25 (21.70)
  Fatigue, 3 months (n=21,33) | 27.78 (23.70) | 43.10 (31.76)
  Fatigue, 6 months (n=20,24) | 36.67 (29.09) | 37.96 (23.61)
  Fatigue, End of Treatment (n=13,24) | 34.19 (28.85) | 34.49 (32.93)
  Nausea and vomiting, Baseline (n=30,42) | 6.67 (14.91) | 2.78 (7.29)
  Nausea and vomiting, 3 months (n=22,33) | 10.61 (14.13) | 9.60 (16.15)
  Nausea and vomiting, 6 months (n=21,24) | 8.73 (17.97) | 7.64 (12.98)
  Nausea and vomiting, End of Treatment (n=13,24) | 10.26 (19.88) | 6.25 (14.59)
  Pain, Baseline (n=30,43) | 14.44 (19.44) | 21.71 (27.83)
  Pain, 3 months (n=22,33) | 12.88 (18.50) | 18.18 (25.47)
  Pain, 6 months (n=21,24) | 23.02 (31.83) | 17.36 (19.95)
  Pain, End of Treatment (n=13,24) | 20.51 (28.18) | 26.39 (32.94)
  Dyspnea, Baseline (n=30,43) | 16.67 (25.89) | 16.28 (25.59)
  Dyspnea, 3 months (n=21,33) | 12.70 (19.65) | 30.30 (32.66)
  Dyspnea, 6 months (n=21,23) | 19.05 (24.88) | 23.19 (29.19)
  Dyspnea, End of Treatment (n=13,24) | 20.51 (28.99) | 23.61 (30.26)
  Insomnia, Baseline (n=30,43) | 24.44 (27.59) | 24.03 (24.48)
  Insomnia, 3 months (n=21,33) | 20.63 (22.30) | 27.27 (30.57)
  Insomnia, 6 months (n=21,24) | 33.33 (34.96) | 29.17 (30.00)
  Insomnia, End of Treatment (n=13,24) | 23.08 (25.04) | 30.56 (33.93)
  Appetite loss, Baseline (n=29,42) | 12.64 (16.46) | 8.73 (20.90)
  Appetite loss, 3 months (n=22,33) | 7.58 (14.30) | 20.20 (24.92)
  Appetite loss, 6 months (n=21,24) | 15.87 (27.12) | 25.00 (26.47)
  Appetite loss, End of Treatment (n=13,24) | 12.82 (28.99) | 25.00 (32.97)
  Constipation, Baseline (n=27,40) | 4.94 (15.20) | 10.00 (21.62)
  Constipation, 3 months (n=21,33) | 15.87 (27.12) | 7.07 (18.18)
  Constipation, 6 months (n=21,23) | 17.46 (27.12) | 11.59 (21.58)
  Constipation, End of Treatment (n=13,24) | 12.82 (21.68) | 13.89 (25.85)
  Diarrhea, Baseline (n=30,41) | 13.33 (24.13) | 37.40 (31.79)
  Diarrhea, 3 months (n=22,32) | 9.09 (21.04) | 45.83 (34.65)
  Diarrhea, 6 months (n=21,23) | 6.35 (17.06) | 43.48 (30.87)
  Diarrhea, End of Treatment (n=12,22) | 2.78 (9.62) | 28.79 (31.36)
  Financial difficulties, Baseline (n=30,413) | 14.44 (25.80) | 8.13 (17.92)
  Financial difficulties, 3 months (n=22,33) | 9.09 (15.19) | 6.06 (15.49)
  Financial difficulties, 6 months (n=21,23) | 15.87 (24.99) | 2.90 (9.60)
  Financial difficulties, End of treatment (n=13,24) | 17.95 (25.88) | 4.17 (14.95)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the date of first dose of study medication until 28 days after the last dose of study medication. Related serious AEs and AEs of special interest (AESIs) were recorded during follow-up.
Description: All participants who received at least 1 dose of study treatment were included in the safety population. A separate analysis of nonserious AEs was not performed, therefore the AEs presented in the other nonserious AE table include all AEs reported during the study, not just nonserious events.
Groups:
- Bevacizumab + Capecitabine: Cycles 1-9 (21-Day cycle): Participants received bevacizumab 7.5 mg/kg IV on Day 1; capecitabine 2000 mg/m^2 tablets PO in a divided dose every 12 hours within 30 minutes following a meal, on Days 1 through 14. Days 15-21 were a rest period. This 21-day cycle was repeated at least 8 times.
Arm/Group | Bevacizumab + 5-FU + Streptozocin | Bevacizumab + Capecitabine
Serious Adverse Events (participants affected / at risk) | 11/34 | 13/49
Other Adverse Events (participants affected / at risk) | 34/34 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + 5-FU + Streptozocin (N=34) | Bevacizumab + Capecitabine (N=49)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
General physical health deterioration (General disorders) | 0 | 2
Influenza like illness (General disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Post-procedural sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Hemorrhage (General disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Thrombotic microangiopathy (Vascular disorders) | 1 | 0
Hemorrhagic stroke (Nervous system disorders) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + 5-FU + Streptozocin (N=34) | Bevacizumab + Capecitabine (N=49)
Nausea (Gastrointestinal disorders) | 24 | 24
Diarrhoea (Gastrointestinal disorders) | 12 | 32
Constipation (Gastrointestinal disorders) | 19 | 9
Abdominal pain (Gastrointestinal disorders) | 13 | 12
Abdominal pain upper (Gastrointestinal disorders) | 11 | 11
Vomiting (Gastrointestinal disorders) | 11 | 7
Haemorrhoids (Gastrointestinal disorders) | 4 | 5
Dry mouth (Gastrointestinal disorders) | 4 | 4
Aphthous stomatitis (Gastrointestinal disorders) | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Flatulence (Gastrointestinal disorders) | 2 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Loose tooth (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Steatorrhoea (Gastrointestinal disorders) | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1
Tongue haematoma (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 23 | 28
Mucosal inflammation (General disorders) | 14 | 17
Oedema peripheral (General disorders) | 4 | 9
Pyrexia (General disorders) | 8 | 4
Fatigue (General disorders) | 4 | 5
Xerosis (General disorders) | 1 | 3
Chest pain (General disorders) | 1 | 2
Chills (General disorders) | 3 | 0
General physical health deterioration (General disorders) | 0 | 3
Influenza like illness (General disorders) | 3 | 0
Malaise (General disorders) | 0 | 2
Oedema (General disorders) | 2 | 0
Catheter site haematoma (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Drug intolerance (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Implant site inflammation (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Mucosal dryness (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 6 | 6
Insomnia (Psychiatric disorders) | 4 | 5
Depression (Psychiatric disorders) | 1 | 3
Confusional state (Psychiatric disorders) | 0 | 3
Sleep disorder (Psychiatric disorders) | 0 | 2
Stress (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 2 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 5
Lymphopenia (Blood and lymphatic system disorders) | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Erosive balanitis (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 2 | 0
Visual impairment (Eye disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea extertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Weight decreased (Investigations) | 4 | 5
Blood bilirubin abnormal (Investigations) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase abnormal (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Haemoglobin (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 2 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 2 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 3
Dysuria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Albuminuria (Renal and urinary disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 13 | 14
Paraesthesia (Nervous system disorders) | 4 | 4
Dizziness (Nervous system disorders) | 3 | 4
Dysgeusia (Nervous system disorders) | 0 | 4
Dysaesthesia (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 1 | 1
Ageusia (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 4
Bronchitis (Infections and infestations) | 3 | 3
Gastroenteritis (Infections and infestations) | 2 | 4
Pharyngitis (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 4
Sinusitis (Infections and infestations) | 2 | 2
Tonsillitis (Infections and infestations) | 3 | 1
Cystitis (Infections and infestations) | 1 | 2
Herpes simplex (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 1 | 2
Oral herpes (Infections and infestations) | 2 | 1
Tooth abscess (Infections and infestations) | 1 | 2
Injection site infection (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 0 | 2
Candidiasis (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Gastroenteritis escherichia coli (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0
Infected cyst (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 | 0
Hyposideraemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 9
Hot flush (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
Vein discolouration (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Bite (Injury, poisoning and procedural complications) | 0 | 1
Burn of internal organs (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Frostbite (Injury, poisoning and procedural complications) | 1 | 0
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Non-obstructive cardiomyopathy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 31
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 8
Erythema (Skin and subcutaneous tissue disorders) | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkeratosis palmaris and plantaris (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discomfort (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Spider naevus (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.